CLINICAL TRIAL: NCT07113093
Title: Effects of Augmented Reality and Virtual Reality-Assisted Gait Training on Balance and Walking in Individuals With Stroke
Brief Title: The Effects of Augmented Reality Versus Virtual Reality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Murat Akıncı, Principal Investigator, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: VR02
Record Dates: First submitted 2025-07-30; First posted 2025-08-08 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: Stroke; Virtual Reality; Augmented Reality; Treadmill
MeSH Terms: conditions — Stroke | interventions — Bro protein, Drosophila

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Augmented Reality (Experimental): In this group, augmented reality will be used during treadmill walking.
  Interventions: Other: Augmented Reality; Other: Others
- Virtual Reality (Experimental): In this group, virtual reality will be used during treadmill walking.
  Interventions: Other: Virtual Reality; Other: Others
- Control Group (Other): Participants in this group will be enrolled in a self-directed exercise program that is matched in duration and content to the VR-AR interventions.
  Interventions: Other: Self Directed Exercises; Other: Others

INTERVENTIONS:
Other: Augmented Reality — Gait training will be conducted using the AR applications Stepping Stones, Reactive Stones, Obstacles, Speed Adjustment, Slalom, Tandem, and Monster Game for 45 minutes.
  Arms: Augmented Reality
Other: Virtual Reality — Gait training will be conducted using the VR applications Nature Island, Italian Apps, and Soccer for 45 minutes.
  Arms: Virtual Reality
Other: Self Directed Exercises — "Patients will be taught exercises including walking on a flat surface, walking with varying step lengths, walking over obstacles, and walking at different speeds. They will be instructed to perform these exercises for 45 minutes per day.
  Arms: Control Group
Other: Others — The treatment duration is 60 minutes. Based on the patient's needs, the following exercises will be performed: scapular and thoracolumbar mobilization; upper and lower extremity exercises (range of motion, stretching, and strengthening); bed mobility and transitional movements such as rolling, coming to a sitting position, and standing up; core activation exercises such as bridging and functional reaching; weight shifting and balance training; gait training (e.g., walking between parallel bars, walking in different directions, and walking over obstacles); and cycling on a bicycle ergometer.

SUMMARY:
This randomized controlled trial aims to compare the effects of augmented reality (AR) and virtual reality (VR)-assisted treadmill gait training on balance and walking in individuals with stroke, within the framework of the International Classification of Functioning, Disability and Health (ICF). A total of 66 post-stroke patients will be randomly assigned to three groups: (1) VR group receiving gait training via C-Mill VR applications in addition to conventional physiotherapy, (2) AR group receiving gait training via C-Mill AR applications in addition to conventional physiotherapy, and (3) control group receiving a home exercise program alongside conventional physiotherapy. Participants will train for 45 minutes per day, five days a week, for three weeks. Outcome measures will include clinical, functional, cognitive, and spatiotemporal gait parameters to evaluate changes in balance and walking ability before and after the intervention.

DETAILED DESCRIPTION:
This prospective, randomized controlled study aims to compare the effects of augmented reality (AR) and virtual reality (VR)-assisted treadmill gait training on balance and walking in individuals with stroke, and to contribute to the literature through a comprehensive analysis within the International Classification of Functioning, Disability and Health (ICF) framework. Stroke is a leading cause of long-term disability and care burden, with nearly one-third of acute stroke survivors unable to walk three months after onset. Improving walking ability is a central goal of stroke rehabilitation. There is increasing evidence that high-intensity, task-specific, and repetitive training can enhance functional recovery. Treadmill training enables intensive, repetitive practice of complex gait patterns and has been shown to improve walking speed and distance in stroke survivors. Technological advances have introduced immersive tools such as VR and AR systems into rehabilitation, providing engaging and interactive environments that enhance motor learning and patient motivation.

The C-Mill VR+ system (Motek, Netherlands) is a treadmill equipped with both AR and VR applications, offering visual-auditory feedback, safety harnesses, and force sensors. Though studies suggest C-Mill training improves gait and reduces fall risk in geriatric and Parkinson's disease populations, comprehensive randomized controlled trials comparing AR- and VR-supported treadmill training in stroke rehabilitation are lacking.

This study will enroll 66 individuals with stroke undergoing inpatient rehabilitation at the Virtual Reality Laboratory of Ankara Bilkent City Hospital. Inclusion criteria include diagnosis of hemiplegia (ICD-10 code G81), age 18 or older, and ability to walk with or without assistance (Functional Ambulation Classification ≥ 2). Exclusion criteria include aphasia, MoCA score <10, additional neurological/orthopedic problems, recurrent stroke, or a Modified Ashworth Scale (MAS) score of 3-4 in the lower extremities. Participants will be randomly assigned to one of three groups: (1) VR group-C-Mill VR treadmill training with Nature Island, Italian Apps, and Soccer applications; (2) AR group-C-Mill AR training using Stepping Stones, Reactive Stones, Obstacles, Speed Adjustment, Slalom, Tandem, and Monster Game applications; (3) Control group-home-based walking exercises (flat ground, variable step length, obstacles, and speed) in addition to standard physiotherapy. All groups will continue routine physiotherapy and receive 45-minute training sessions, five days a week for three weeks.

Outcome measures assessed pre- and post-intervention include the Timed Up and Go Test, Fugl-Meyer Lower Extremity Motor Assessment, Modified Ashworth Scale, Activities-specific Balance Confidence Scale, Berg Balance Scale, Functional Ambulation Classification, Trunk Impairment Scale, Stroke Impact Scale (3.0), Stroke-Specific Quality of Life Scale, Montreal Cognitive Assessment (MoCA), and spatiotemporal gait analysis via the C-Mill VR+ system. Gait analysis will record step lengths, stance and swing phases, and double support percentages for both paretic and non-paretic limbs at self-selected and fixed speeds.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 diagnosis code of G.81 (Hemiplegia)
* Age 18 years or older
* Ability to walk with assistance or independently (Functional Ambulation Classification score of 2 or higher)

Exclusion Criteria:

* Incomplete completion of the assessment form
* Refusal to participate in the study
* Aphasia
* Montreal Cognitive Assessment score below 10
* Presence of extra neurological or orthopedic problems unrelated to stroke
* Recurrent stroke
* MAS score of 3-4 (lower extremity)
* Volunteer's desire to withdraw from the study
* Inability to adapt to the technological devices used in the study (e.g., visual or hearing impairments)
* Missing three consecutive treatment sessions
* Botulinum toxin-A (BONT-A) injection to the lower extremity during the treatment process or within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) Test | baseline and after 3 weeks
  To perform the test, the patient stands up from a chair approximately 46 cm in height, walks at a comfortable and safe pace to a marked target three meters away, turns around the target, and returns to sit back down on the chair. To ensure familiarity with the procedure, the patient performs one trial without timing. If needed, the patient may use their usual walking aid (e.g., cane or walker). A shorter completion time indicates better performance.
Berg Balance Scale (BBS) | baseline and after 3 weeks
  The scale consists of 14 items and assesses the patient's ability to maintain balance (either static or during various functional movements) over a specific period of time. Each item is scored on a scale from 0 to 4:
  0 points: Unable to complete the task. 4 points: Completes the task independently. The maximum total score is 56. A score of 0-20 indicates poor balance, 21-40 indicates acceptable balance, and 41-56 indicates good balance.
Gait Analsis | baseline and after 3 weeks
  Spatio-temporal gait analysis will be performed using the C-Mill VR+ device. As a result of this measurement, step lengths, stance phases (%), swing phases (%), and double support phases (%) of the paretic and non-paretic limbs will be recorded. Gait analysis will be conducted in two separate assessments: at the participant's self-selected comfortable walking speed and at a fixed speed of 1 km/h. The gait analysis will begin after a 2-minute warm-up period, and data will be collected for the following 2 minutes. A rest period of at least 5 minutes will be provided between the two assessments.

SECONDARY OUTCOMES:
Fugl-Meyer Motor Assessment Lower Extremity (FMA-LE) | baseline and after 3 weeks
  The FMA is a widely used, valid, and reliable test for evaluating motor impairments of the paretic upper and lower extremities in stroke patients. Each item on the scale is scored as follows: 0 = unable to perform, 1 = performs partially, and 2 = performs fully. Higher scores indicate better motor function. In this study, the 34-point lower extremity section of the scale will be used.
Activities-specific Balance Confidence (ABC) Scale | baseline and after 3 weeks
  The ABC Scale is a 16-item self-assessment questionnaire that asks individuals to rate their confidence in maintaining balance during specific ambulatory activities on a numerical scale from 0 to 100. A score of 0 represents no confidence at all, while a score of 100 represents complete confidence in performing the activity. Each participant's total ABC score is calculated by summing the scores for each item and then dividing by the number of items. Botner et al. reported that the scale can be used to assess fear of falling in individuals with stroke. Myers and colleagues suggested that ABC scores below 50 indicate low physical function, scores between 50 and 80 indicate moderate physical function, and scores above 80 indicate high functionality among physically active older adults.
Functional Ambulation Category (FAC) | baseline and after 3 weeks
  The FAC is a valid and reliable scale used in patients with post-stroke hemiparesis that classifies walking ability into six levels based on the amount of physical assistance required. A score of 0 indicates that the patient needs assistance from two people to walk, while a score of 5 represents independent walking on all surfaces including stairs.
Trunk Impairment Scale (TIS) | baseline and after 3 weeks
  The scale was developed to assess trunk function after stroke. It consists of three sections: static sitting balance, dynamic sitting balance, and coordination. Due to a ceiling effect in the static sitting balance section, a revised version was developed in 2010 that excludes this section. This new version is recommended for patients with mild to moderate impairment and those in the chronic phase.
Stroke Impact Scale (SIS) Version 3.0 | baseline and after 3 weeks
  The SIS is a comprehensive health status measure specifically designed for stroke. It consists of 8 domains and 59 items. Each item is rated on a scale from 1 to 5. For items 3f, 3h, and 3i in domain 3, reverse scoring is applied using the formula (6 - the marked score). A new domain has been added to assess the patient's overall perception of recovery, where the patient rates their recovery on a scale from 0 to 100. The score for each subdomain is calculated using the formula:
  Subdomain Score = ((Mean Item Score - 1) / 4) × 100
Stroke-Specific Quality of Life Scale (SS-QOL) | baseline and after 3 weeks
  The scale consists of 12 domains-Thinking, Personality, Mood, Family Roles, Social Roles, Energy, Self-Care, Vision, Language, Mobility, Work/Productivity, and Upper Extremity Function-and includes a total of 49 items. Each item is scored using a 5-point Likert scale based on the patient's experience during the past week. The overall quality of life score is the sum of the scores from all subdomains. Higher scores indicate better quality of life. Subdomains can also be analyzed independently to identify specific areas of difficulty.

OTHER OUTCOMES:
Modified Ashworth Scale (MAS) | baseline and after 3 weeks
  For the soleus muscle, the patient is positioned in a side-lying posture with the hips flexed at 45° and the knees flexed at 45°. For the gastrocnemius muscle, the patient remains in side-lying position with hips flexed at 45° and knees fully extended. The head and trunk are aligned in a straight line. The evaluator, positioned in front of the patient, stabilizes the lower leg proximally at the ankle joint with one hand, while the other hand is placed under the foot. The thumb is placed on the lateral surface of the calcaneus, fingers on the medial surface, and the palm supports the sole of the foot. The patient is instructed to relax as much as possible. The ankle is moved from maximum plantarflexion to maximum dorsiflexion.
  For the quadriceps femoris muscle, the patient lies in side-lying position with hips and knees fully extended. The evaluator stands behind the patient, stabilizes the thigh proximally near the knee on the lateral surface with one hand, and places the other hand
Montreal Cognitive Assessment (MoCA) | baseline and after 3 weeks
  The MoCA is a valid screening test designed for the rapid assessment of mild cognitive impairment in individuals post-stroke. It is a one-page, 30-point test that evaluates various cognitive domains including visuospatial abilities, executive functions, short-term memory, attention, language, and orientation to time and place. Scores of 26 and above are generally considered normal, 18-25 indicate Mild Cognitive Impairment, 10-17 suggest Moderate Dementia, and scores below 10 indicate Severe Dementia. An adjustment of +1 point can be made for individuals with lower education levels (12 years or less of formal education).

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided